CLINICAL TRIAL: NCT02875002
Title: Phase 1 Study of Volasertib and Belinostat in Patients With Relapsed and Refractory Aggressive B-cell and T-cell Lymphomas
Brief Title: Study of Volasertib and Belinostat in Patients With Relapsed and Refractory Aggressive B-cell and T-cell Lymphomas
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Massey Cancer Center (Other); Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1601017105
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Relapsed and Refractory Aggressive B- and T-cell Lymphomas; Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, T-Cell; Lymphoma | interventions — BI 6727; belinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Experimental): Subjects have relapsed and refractory aggressive B- and T-cell lymphomas and will receive both Belinostat and Volasertib.
  Interventions: Drug: volasertib; Drug: belinostat

INTERVENTIONS:
Drug: volasertib — Volasertib (BI6727) is a small molecule inhibitor of the polo-like kinase 1 (PLK1) protein. Infusion for 60 minutes. Dosing will start at 25 mg/m^2, is schedule to increase to 100mg/m^2, and be administered on days 1 and 8 of each 28-day cycle.
Drug: belinostat — Belinostat is a histone deacetylase inhibitor. Infusion will take 30 minutes. Dosing will start at 600 mg/m^2 , is scheduled to increase to 1000 mg/m^2, and will be administered on days 1,2,3 and 8,9,10 of each 28-day cycle.

SUMMARY:
This phase 1, multicenter, open-label study is designed to find the RP2D of volasertib, a PLK1 inhibitor, and belinostat, an HDAC inhibitor, when given in combination to patients with relapsed or refractory B-cell or T-cell lymphoma. A standard 3+3 dose-escalation design will be employed with study enrollment beginning at dose level 1.

ELIGIBILITY:
Inclusion Criteria:

A patient must meet all of the following inclusion criteria to be eligible to participate in the study.

* Histologically confirmed aggressive B-cell or T-cell lymphoma including the following:
* B-cell lymphomas
* DLBCL (including transformed follicular lymphoma)
* Mantle cell lymphoma
* Burkitt lymphoma
* Peripheral T-cell lymphoma (PTCL) excluding cutaneous T-cell lymphoma
* Disease that is relapsed or refractory after a minimum of 2 previous therapies, if B-cell lymphoma, or a minimum of 1 previous therapy, if PTCL
* For patients who have had autologous stem cell transplant, disease relapse must be more than 100 days following transplant.
* For patients who have had allogeneic stem cell transplant, all of the following conditions must be met:
* ≥ 6 months since allogeneic transplant
* Graft vs. host disease (GVHD) is not present
* Patient is not currently on immunosuppressive therapy
* At least one site of measurable disease by PET/CT: a node measurable in 2 diameters and with longest diameter >1.5cm or an extranodal lesion measurable in 2 diameters and with longest diameter >1cm.
* Age ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 (see Appendix 1)
* Life expectancy of at least 3 months
* CBC with differential providing evidence of adequate bone marrow function as defined below:
* Absolute neutrophil count (ANC) ≥ 1500/mm3 without growth factor support for 7 days
* Platelets ≥ 75,000/mm3 (without transfusion for 7 days)
* Adequate renal function defined as: Creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated or actual creatinine clearance ≥ 60 mL/min (see Appendix 2 for the Cockcroft -Gault Formula to calculate creatinine clearance)
* Adequate hepatic function as defined below:
* AST ≤ 2.5 x ULN
* ALT ≤ 2.5 x ULN
* Total bilirubin ≤ 1.5 mg/dL
* Note: Patients with documented Gilbert's syndrome are eligible if total bilirubin is ≤ 3.0 mg/dL.
* Serum potassium and serum magnesium within normal limits Note: Electrolytes may be corrected with supplementation.
* For a woman of childbearing potential (WCBP), a negative serum pregnancy test performed within 14 days prior to study enrollment (7 days prior to initiation of study treatment) Note: WCBP is defined as any woman who has not had a hysterectomy or bilateral oophorectomy and is not postmenopausal (i.e., she has had menses in the preceding 24 consecutive months)
* WCBP and male patients must agree to use a highly effective method of birth control for the duration of study treatment and for 6 months following completion of study treatment Note: A highly effective method of contraception is defined as one that results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomised partner.
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

A patient who meets any of the following exclusion criteria is ineligible to participate in the study.

* Any investigational treatment within 30 days prior to initiation of study treatment
* Plans for concurrent treatment with other investigational agents
* Plans for other concurrent cancer treatment including steroids for cancer control
* Chemotherapy or large field radiotherapy within 3 weeks prior to initiation of study treatment
* Previous histone deacetylase inhibitor administered as cancer treatment.
* History of brain metastasis including leptomeningeal metastasis
* QTc interval ≥450 (i.e., ≥ grade 0, per CTCAE version 4) on ECG prior to initiation of study treatment. If baseline QTc on screening ECG is ≥ 450 ms (i.e., ≥ grade 1)
* Check potassium and magnesium serum levels
* Correct any identified hypokalemia and/or hypomagnesemia and repeat ECG to confirm QTc interval
* For patients with baseline HR < 60 or > 100 bpm, manual read of QT by cardiologist is required, with Fridericia correction applied to determine the QTcF interval.
* Note: For patients with HR 60-100 bpm, no manual read of QTc is required.
* Any of the following related to risk of torsades de pointes and sudden cardiac death:
* History of sustained ventricular tachycardia (VT, ventricular fibrillation (VF), torsades de pointes, or resuscitated cardiac arrest unless currently addressed with an implanted cardiac defibrillator
* Concomitant treatment with an anti-arrhythmic agent to prevent or control arrhythmia. Agents used for rate-control of atrial fibrillation are permitted provide that they are not prohibited due to potential drug interactions (see Section 6.4)
* Known congenital long QT syndrome
* Second degree atrioventricular (AV) block type II, third degree AV block, or ventricular rate < 50 bpm
* Any of the following related to ischemic heart disease:
* Angina with ordinary physical activity
* Note: If angina only occurs with strenuous, rapid, or prolonged exertion, the patient is eligible.
* Myocardial infarction within 6 months prior to study enrollment
* Note: If myocardial infarction occurred within 6-12 months prior to study enrollment, patient must be asymptomatic and have had a negative cardiac risk assessment (e.g., treadmill stress test, nuclear medicine stress test, or stress echocardiogram)
* ECG with evidence of cardiac ischemia (i.e., ST depression of ≥ 2 mm, measured from isoelectric line to ST segment; T-wave inversion ≥ 4 mm measured from isoelectric line to peak of T-wave)
* Any of the following related to heart failure:
* New York Heart Association (NYHA) class II, III or IV congestive heart failure (see Appendix 3) or known left ventricular ejection fraction < 40% by MUGA scan or < 50% by echocardiogram or MRI
* Known hypertrophic cardiomegaly or restrictive cardiomyopathy
* Clinically significant infection including active hepatitis B or hepatitis C requiring treatment
* Known human immunodeficiency virus (HIV) seropositivity nNote: HIV testing is not required
* History of allergic reactions attributed to compounds similar to the chemical or biologic composition of belinostat or volasertib
* History of another primary malignancy, excluding non-melanoma skin cancer, cervical carcinoma in situ, and/or other in situ cancers treated by local excision, that has not been in remission for at least 2 years
* Pregnancy or breastfeeding
* Medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk, interfere with the patient's participation in the study, or hinder evaluation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2018-03 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Doses (MTD) | up to 2 years
  Dose escalation will follow the traditional 3+3 plan to determine the MTD and the recommended phase 2 doses (RP2D). The MTD will be defined as that dose level at which ≤ 1/6 patients experience Dose Limited Toxicity (DLT), with ≥ 2/6 experiencing DLT at the next higher dose level.
  If the MTD is not reached at dose level 5, consideration will be given to amending the dose level escalation schema to add an additional dose level.
Adverse Events | up to 2 years
  To evaluate the safety and toxicity of volasertib and belinostat when given in combination

CONTACTS AND LOCATIONS:
Overall Officials: Steven Gore, MD, Principal Investigator — Yale University; Iris Isufi, MD, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Yale Cancer Center, New Haven, Connecticut
  - Sidney Kimmel Comprehensive Cancer, Baltimore, Maryland
  - Massey Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No